CLINICAL TRIAL: NCT05724043
Title: Assessment of the SmartJournal Intervention for Improved Oral Care in Nursing Homes: an Evaluation Study
Brief Title: SmartJournal for Improved Oral Care in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oral Health Center of Expertise Rogaland, Norway (Other)
Collaborators: University of Bergen (Other); University of Stavanger (Other); Regional Research Funds Rogaland, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REK 2022/472796
Record Dates: First submitted 2023-01-10; First posted 2023-02-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Oral Health
Keywords: Oral health; Care-dependent elderly; Nursing home; Nursing staff; Intervention; Digital tool

STUDY DESIGN:
Intervention Model Description: A pragmatic cluster randomized controlled trial (C-RCT) will be employed to assess effects of SmartJournal usage as specified in the study objectives. Nursing homes located in Rogaland, Norway, will be recruited and randomly assigned to an intervention group and a control group. Nursing homes in the intervention group will be provided with tablets containing SmartJournal and receive training and follow-up throughout the intervention period. Nursing homes in the control group will continue with existing oral care routines. The intervention will last for 12 weeks.
Who Masked: Participant, Care Provider
Masking Description: Participants will not receive information about who is included in the intervention- and control group, respectively. They will only receive information that is relevant for their participation. The chosen study design (C-RCT) facilitates this masking by reducing the possibility of contamination between the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmartJournal (Experimental): Nursing homes in the intervention group will receive the SmartJournal intervention. They will be provided with toolboxes including tablets with SmartJournal installed, antibacterial touchscreen wipes, flashlights for monthly oral inspections, instruction video, instruction book and SmartJournal information posters. They will also receive oral hygiene equipment packages including toothbrushes for permanent teeth and prosthetic devices, dental floss, interdental brushes, toothpaste and inspection mirrors. Training, follow-up and technical support for SmartJournal usage will be provided by project staff employed at the Oral Health Centre of Expertise Rogaland. The intervention will last for 12 weeks.
  Interventions: Device: SmartJournal
- Control group (No Intervention): Nursing homes in the control group will also receive oral hygiene equipment packages but will, in contrast to the intervention group, continue with existing oral care routines.

INTERVENTIONS:
Device: SmartJournal — SmartJournal is a tablet application with three modules: Module 1 offers a system for simple check-box registration of daily oral hygiene routines. This module also includes an open text field where the caregiver can give a brief description of strategies used if the patient shows resistant behaviors. Module 2 offers a system for monitoring the patient's oral health through monthly check-ups. This module is an image-based, interactive learning- and assessment tool. Upon completion of the monthly oral health assessment health personnel receive a summary report with suggestions for tailored preventive and/or curative measures to be initiated. Module 3 offers an easily accessible knowledge base which includes information on geriatric oral health, standard equipment and procedures for daily oral hygiene routines for patients with various care needs. It also includes scientifically documented strategies that may be used to approach patients with dementia refusing oral care assistance.
  Arms: SmartJournal

SUMMARY:
Poor oral health is common in care-dependent older adults, and healthcare professionals report numerous barriers when it comes to provision of oral care for elderly patients. Frequently reported barriers are lack of oral health knowledge/skills and care resistant behaviors (CRB) in patients suffering from dementia. Other barriers include lack of adequate oral care routines and satisfactory systems for documentation of issues related to oral health, a high workload and unclear responsibilities. To overcome these barriers, an easy-to-use digital tool named SmartJournal has been developed to assist health personnel in preserving the older patient's oral health. SmartJournal has three components: one for documentation of oral hygiene routines, one for monthly oral health assessment and one for e-learning (a digital knowledge base with information on geriatric oral health and handling of CRB). The objectives of the present study are to assess: 1) the effectiveness of SmartJournal in enhancing nursing home caregivers' capability, opportunity, motivation and routines related to oral care, 2) whether SmartJournal usage may result in improved oral health for nursing home residents and 3) whether SmartJournal usage may result in changes in documentation of oral health related issues in patient journals.

A cluster randomized controlled trial (C-RCT) will be employed to assess effects of SmartJournal usage as specified in the study objectives. Nursing homes located in Rogaland, Norway, will be recruited and randomly assigned to an intervention- and a control group. The intervention group will be provided with tablets containing SmartJournal, while the control group will continue with existing oral care routines. The intervention will last for 12 weeks. Measurements will be performed in both groups at baseline, immediately post-intervention (3 months) and at follow-up (9 months) and include: 1) a survey assessing caregivers' capability, opportunity, motivation and routines related to oral care, 2) oral examinations in residents using mucosal-plaque score (MPS) as a primary outcome variable for assessing oral health status, and 3) examination of patient journals to assess the frequency and quality of reported oral health related issues. We hypothesize that SmartJournal usage will have a positive effect as measured by favorable changes in study variable scores.

DETAILED DESCRIPTION:
INTRODUCTION

Poor oral health is common in frail and care-dependent older adults and includes tooth loss, poor oral hygiene, high prevalence of dental caries and periodontal disease, defective dental prostheses, hyposalivation and various oral lesions caused by misfitting dentures and/or precancerous or cancerous states. Alarmingly, oral health is shown to be the most neglected area in Norwegian nursing homes and oral healthcare is the first task to be downgraded due to lack of resources. Neglect of oral health, resulting in poor oral hygiene, may cause infections and inflammation both locally and systemically. Oral infections have been associated with systemic conditions such as atherosclerosis, diabetes and aspiration pneumonia. Moreover, chewing difficulties as a result of poor dental status have been associated with altered dietary habits, malnutrition and cognitive decline. According to the World Health Organization, this is a worldwide problem as oral health is an often neglected area of healthy ageing. A few decades ago, most older adults were denture wearers. Today, an increasing number of elderly keep their natural teeth - often in combination with complex and expensive fixed and/or removable prosthesis. While dentures are easy to manage, the more complex prosthetic devices can represent a challenge with regard to handling and cleaning. Thus, care-dependent elderly have to rely on caregivers to maintain satisfactory oral health. Research from Sweden and Denmark has shown that about 80% of nursing home residents need assistance with daily oral hygiene practices. Thus, it is disturbing that healthcare professionals report numerous barriers when it comes to provision of adequate oral care. The most frequently reported barriers are lack of knowledge and skills and care resistant behaviors (CRB), in particular among patients suffering from dementia. Research has indicated that more than 50% of Norwegian nursing home residents with dementia refuse oral care assistance. In cases of frequent CRB, daily oral care may be postponed repeatedly, resulting in poor oral hygiene and increased risk of oral and systemic infections. Other reported barriers include lack of adequate oral care routines, lack of systems for documentation of issues related to oral health, a high workload and unclear responsibilities. To overcome the reported barriers for provision of adequate oral care in the elderly, an interactive and easy-to-use digital tool named SmartJournal has been developed to assist health personnel in preserving nursing home residents' oral health. SmartJournal, which is an application for tablet, is created by researchers at the Oral Health Centre of Expertise in Rogaland, Norway, in close collaboration with dental professionals, nursing home caregivers and innovative research- and development environments. The objectives of the current research are: to assess 1) the effectiveness of SmartJournal in enhancing nursing home caregivers' capability, opportunity, motivation and routines related to oral care, 2) whether SmartJournal usage may result in improved oral health for nursing home residents and 3) whether SmartJournal usage may result in changes in the documentation of oral health related issues in patient journals.

METHODS

Design and procedures

A pragmatic cluster randomized controlled trial (C-RCT) will be employed to assess effects of SmartJournal usage as specified in the study objectives. Nursing homes located in Rogaland, Norway, will be recruited and randomly assigned to an intervention group and a control group. Nursing homes in the intervention group will be provided with tablets containing SmartJournal, while nursing homes in the control group will continue with existing oral care routines. The intervention will last for 12 weeks. Following recruitment of participants and baseline measurements, nursing homes in the intervention group will be provided with SmartJournal toolboxes and packages with oral hygiene equipment, while nursing homes in the control group will receive oral hygiene equipment packages only. Training, follow-up and technical support for SmartJournal users will be provided by project staff employed at the Oral Health Centre of Expertise Rogaland.

Measurements

Effects of SmartJournal usage on caregivers' capability, opportunity, motivation and routines related to oral healthcare and handling of CRB will be measured by a survey questionnaire. Caregivers in both the intervention- and the control group will be asked to fill out the survey questionnaire three times: before the intervention (baseline), immediately after the intervention (at 3 months) and 6 months after the intervention (at 9 months). Effects of SmartJournal usage on nursing home residents' oral health will be assessed using the mucosal-plaque score (MPS) as a primary outcome measure. Residents in both the intervention- and the control group will have an assessment of MPS at three times: at baseline, 3 months and 9 months. MPS assessments will be performed by dental professionals employed at the Oral Health Center of Expertise Rogaland, Norway. Calibration will be undertaken to ensure reliability of the clinical measurements. Effects of SmartJournal usage on documentation of oral health related issues in patient journals will be measured both quantitatively (i.e., frequency of documentation) and qualitatively (i.e., qualitative assessment of documentation) at three times throughout the project period: at baseline, 3 months and 9 months. Additional journal data shown to be associated with oral health will also be retrieved and used to describe the study sample and to be included as covariates in statistical analyses. These data include socio-demographics, medical conditions and prescribed medication.

Power and sample size

Estimation of sample size is based on previous research using MPS as a primary outcome measure. We assume an alpha of 0.5, a power of 80% and a 33% drop-out rate due to the residents' frail condition and a median resident time of two years. A medical statistician has been consulted to further adapt the calculations to the present study setting (taking into account the number of eligible nursing homes and residents in Rogaland), recommending the inclusion of 12 nursing homes each with 30 residents opted for oral health assessments. Thus, a total of 360 residents will be included for oral health assessments, 180 in the intervention and control group, respectively. All eligible caregivers in the included nursing homes will be invited to take part in the survey.

Data analyses

The statistical software package SPSS (IBM) will be used for analyses of quantitative data such as survey data, MPS data and frequency data from patient journals. The analyses will include descriptive statistics and statistical techniques to look for changes and differences in the study variables within and between the intervention- and the control group throughout the project period (e.g., t-tests and analysis of variance tests). We hypothesize that SmartJournal usage will lead to favorable changes in variable scores. In caregivers: improved capability, opportunity, motivation and routines related to oral care (survey data). In residents: improved oral health as measured by MPS. In patient journals: enhanced reporting of oral health related issues. Additionally, regression analysis will be employed to investigate associations between study variables while adjusting for potential covariates. NVivo (Alfasoft) will be used to analyze qualitative data from patient journals.

ELIGIBILITY:
INCLUSION CRITERIA

Nursing homes:

* Located in Rogaland county, Norway
* Long-term facilities

Residents (patients):

* Long-term residents (i.e., residents with the nursing home as their permanent address)
* Residents with and without dementia, who can undergo oral examination

Nursing staff:

* All types of nursing staff (nurses, auxiliary nurses, students)
* Full- and parttime staff

EXCLUSION CRITERIA

Nursing homes:

* Specialized nursing homes (e.g., psychiatry, substance abuse)
* Short-term facilities (e.g., rehabilitation, respite care)
* Nursing homes already following a specific protocol for oral care and/or participate in other comprehensive interventions

Residents (patients):

* Short-term residents
* Critically ill and terminal patients receiving palliative care

Nursing staff:

• Staff with purely administrative tasks (e.g., heads of institutions)

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Mucosal-plaque index (MPS) | Change in MPS from baseline at 3 months and 9 at months.
  The primary outcome measure is MPS. MPS is comprised of a four-point plaque score (PS) and a four-point mucosal score (MS). PS = 1: no visible plaque, PS = 2: plaque is barely visible, PS = 3: moderate amount of plaque, PS = 4: large amount of plaque almost covering the whole surface of teeth. MS = 1: normal mucosa, MS = 2: mild inflammation, MS = 3: medium inflammation, MS = 4: strong inflammation. For both scores, if in doubt between 1 and 2, dental personnel are instructed to score 1. If in doubt between 3 and 4, they are instructed to score 4. The index is designed to evaluate oral health and oral hygiene in groups of individuals. This makes it a suitable index to be used when conditions are not optimal to assess the patient's oral health. In a nursing home setting, dental personnel have limited equipment and poor light compared to an ordinary dental clinic setting. Therefore, using an index designed to be applied outside a dental clinic setting is feasible in this research.

SECONDARY OUTCOMES:
Survey data | Change in variable scores for capability, opportunity, motivation and routines (measured in questionnaire) from baseline at 3 months and at 9 months.
  The secondary outcome measure is caregivers' response to a survey assessing effects on identified barriers related to provision of adequate oral care (i.e., a health personnel/caregiver perspective). The survey is designed to measure nursing home caregivers' capability, opportunity, motivation and routines related to oral care. These variables are measured by multiple items with response alternatives on a five-point Likert scale ranging from 'totally disagree' (1) to 'totally agree' (5). Higher scores mean better perceived capability, opportunity, motivation and routines related to oral care.

OTHER OUTCOMES:
Patient journals | For oral health related documentation: change in frequency and content from baseline at 3 months and at 9 months. For sociodemographics, medical conditions and prescribed medication: measurement at baseline only.
  Other pre-specified outcomes include data from patient journals. Journal data include assessment of oral health related documentation, sociodemographics, medical conditions and prescribed medication.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Lind Melbye, PhD, Principal Investigator — Oral Health Centre of Expertise Rogaland, Norway
Locations (1):
- Oral Health Centre of Expertise Rogaland, Norway, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No
IPD from this study will not be shared with researchers outside the project group. This is emphasized in the information- and consent form that will be handed out to potential participants before data collection.

REFERENCES:
- [Derived] Karamehmedovic E, Myhren LE, Jensen KHM, Rodakowska EJ, Astrom AN, Melbye EL. Evaluating the role of the smartjournal digital intervention in improving oral hygiene among nursing home residents: a cluster randomised trial. BMC Oral Health. 2025 Oct 10;25(1):1589. doi: 10.1186/s12903-025-06994-0. PMID 41073970
- [Derived] Melbye EL, Bull VH, Hidle KS. Assessment of the SmartJournal Intervention for Improved Oral Care in Nursing Homes: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2023 Oct 6;12:e46926. doi: 10.2196/46926. PMID 37801358

DOCUMENTS (1):
  • Study Protocol (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT05724043/Prot_000.pdf